CLINICAL TRIAL: NCT01763021
Title: An Open-Label, Sequential Design Study to Assess the Effect of Rifampin on the Pharmacokinetics of PCI-32765 in Healthy Subjects
Brief Title: A Study to Assess the Effect of Rifampin on the Pharmacokinetics of PCI-32765 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR100929; PCI-32765CLL1010 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2013-01-04; First posted 2013-01-08 (Estimated); Last update posted 2013-04-17 (Estimated); Status verified 2013-04

CONDITIONS: Healthy Participants
Keywords: Healthy participants; PCI-32765; Rifampin; PCI-45227; CYP3A4
MeSH Terms: interventions — ibrutinib; Rifampin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PCI-32765 + Rifampin (Experimental): Participants will recieve a single oral dose of PCI-32765 560 mg on Day 1 and Day 11 along with rifampin; and rifampin 600 mg from Day 4 to Day 13.
  Interventions: Drug: PCI-32765; Drug: Rifampin

INTERVENTIONS:
Drug: PCI-32765 — PCI-32765 will be administered as a single oral dose of PCI-32765 560 mg on Day 1 and Day 11
Drug: Rifampin — Rifampin 600 mg (2 X 300 mg) daily dose will be administered orally from Day 4 to Day 13 and on Day 11 along with PCI-32765.

SUMMARY:
The purpose of this study is to assess the potential effects of rifampin on the pharmacokinetics (how the drug concentrations change over time) of PCI-32765 in healthy participants.

DETAILED DESCRIPTION:
This is an open-label (all people know the identity of the intervention), single center (study conducted at one site), sequential study (it is a design in a single group of participants are administered one or more study medication in a sequence) to evaluate the potential effects of rifampin on the pharmacokinetics of PCI-32765 in healthy participants.The study consists of 3 phases: screening phase (21 days prior to first dose of study medication), treatment phase (14 days), and a follow up phase (10 to 12 days after the last dose of study medication). In the treatment phase, a single dose of PCI-32765 560 mg will be administered orally on Day 1 and Day 11. Rifampin 600 mg (2 X 300 mg) will be administered orally on Days 4 to 13; followed by a single dose of PCI-32765 on Day 11. Follow up will be continued until Day 14. Safety evaluations for adverse events, clinical laboratory tests, electrocardiogram, vital signs, and physical examination will be monitored throughout the study. The duration of the study will be approximately for 45 days.

ELIGIBILITY:
Inclusion Criteria:

* Participants should be healthy on the basis of physical examination, medical history, vital signs, electrocardiogram, the results of blood biochemistry and hematology tests and a urinalysis performed at screening
* Agrees to protocol-defined use of effective contraception

Exclusion Criteria:

* Participants with medically significant cardiac disease, hematologic, lipid abnormalities, significant pulmonary disease (bronchospastic respiratory), diabetes mellitus, renal or hepatic insufficiency, thyroid disease, neurologic or psychiatric disease and infectious disease
* Abnormal clinical laboratory and physical examination and vital signs
* Use of any prescription or nonprescription medication (including vitamins and herbal supplements), except for acetaminophen, within 3 days before the first dose of the study drug is scheduled
* Positive to human immunodeficiency virus-type 1 (HIV-1) or HIV-2 test and hepatitis A, B or C infection at screening

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2012-12; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma concentration of PCI-32765 | Day 1 (Predose, 30 minutes, 1, 1.5, 2, 3, 4, 6, 8, 12, and 16 hours), Day 2, Day 3, Day 4, Day 11 (Predose, 30 minutes, 1, 1.5, 2, 3, 4, 6, 8, 12, and 16 hours), Day 12, Day 13 and Day 14
Area under the plasma concentration-time curve from time 0 to time of the last quantifiable concentration of PCI-32765 | Day 1 (Predose, 30 minutes, 1, 1.5, 2, 3, 4, 6, 8, 12, and 16 hours), Day 2, Day 3, Day 4, Day 11 (Predose, 30 minutes, 1, 1.5, 2, 3, 4, 6, 8, 12, and 16 hours), Day 12, Day 13 and Day 14
Area under the plasma concentration-time curve from time 0 to infinite time of PCI-32765 | Day 1 (Predose, 30 minutes, 1, 1.5, 2, 3, 4, 6, 8, 12, and 16 hours), Day 2, Day 3, Day 4, Day 11 (Predose, 30 minutes, 1, 1.5, 2, 3, 4, 6, 8, 12, and 16 hours), Day 12, Day 13 and Day 14

SECONDARY OUTCOMES:
Obsreved plasma concentrations of metabolite PCI-45227 | Day 1 (Predose, 30 minutes, 1, 1.5, 2, 3, 4, 6, 8, 12, and 16 hours), Day 2, Day 3, Day 4, Day 11 (Predose, 30 minutes, 1, 1.5, 2, 3, 4, 6, 8, 12, and 16 hours), Day 12, Day 13 and Day 14
Number of participants with adverse events | up to 45 days

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Neptune City, New Jersey, United States